CLINICAL TRIAL: NCT01467856
Title: Sleep Disordered Breathing (SDB) in Persons With Chronic Tetraplegia: Characterization and Treatment
Brief Title: Sleep Disordered Breathing
Acronym: SDB
Status: Completed | Type: Observational
Sponsor: Mark S. Nash, Ph.D., FACSM (Other)
Responsible Party: Sponsor-Investigator, Mark S. Nash, Ph.D., FACSM, Mark S. Nash, Ph.D., Prinicpal Investigator, University of Miami
Organization: University of Miami (Other)
Other Study IDs: TMP-MN-010
Record Dates: First submitted 2011-09-27; First posted 2011-11-09 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Sleep Disordered Breathing; Tetraplegia
Keywords: Tetraplegia
MeSH Terms: conditions — Sleep Apnea Syndromes; Quadriplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Insulin Sensitivity (SI) and Lipid/Inflammation panels: (30 minutes, Taken at Baseline, 1 month, and 3 month time points) SI will be calculated using the Quantitative Insulin Sensitivity Check Index (QUICKI) method177 that requires single fasting blood glucose and insulin values. The same blood sample will be used to assay for a lipid panel containing total cholesterol, LDL, HDL, and triglycerides and an inflammatory panel testing hs-CRP and IL-6.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic tetraplegia
  Interventions: Procedure: PAP Device Procedure

INTERVENTIONS:
Procedure: PAP Device Procedure — Following titration, subjects will be issued a PAP machine programmed at this optimum pressure and instructed to use the device nightly for the ensuing three months. Compliance checks will be conducted at months 1 and 3 by having the subjects present the PAP "Smartcard" for download and interpretation.
  Daily compliance will be reported as the total number of hours of PAP use per 24 hour period. Patients who use PAP > 4 hours/ night for more than 50% of the nights at one month and 3 month follow-up will be classified as 'compliant' with PAP. Non-compliance will be addressed by a clinical problem-solving approach normally utilized by sleep laboratory personnel in the UM PAP clinic.

SUMMARY:
Sleep-disordered breathing (SDB) occurs in 2% to 4% of the non-disabled adult population and is characterized by periods of complete breathing cessation (apnea) or marked reductions in airflow (hypopnea) during sleep. By contrast, the diagnosis of SDB affects as many as 83% of persons with tetraplegia within one year of their injury. While some consider daytime somnolescence from poor sleep quality a 'tolerable annoyance', SDB can decrease near-term physical performance and mental alertness, decay memory and intellectual processing, invoke mood disturbances, decrease healthrelated quality of life(HRQoL), and cause vehicular or occupational injury. Recurrent sleep arousal is now strongly associated with cardiometabolic (CM) component risks including insulin resistance, obesity, inflammatory stress, and endothelial dysfunction. Despite considerable advancements in understanding and treating SDB - including favored use of positive airway pressure (PAP) - an evidence base sufficient to warrant routine evaluation and treatment of SDB and related sleep disorders remains elusive for those with spinal cord injury (SCI). To address these knowledge and treatment shortcomings the investigators will conduct a hypothesis-driven study with specific aims that will: 1) describe by stakeholder survey the clinically-relevant determinants of sleep quality in persons with chronic tetraplegia, 2) assess clinical features and co-morbid risks associated with SDB in persons with tetraplegia, and 3) determine in persons with tetraplegia having SDB whether treatment using PAP reduces health risks and improves HRQoL. Hypothesis 1 will be tested using data derived from a website survey.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will consecutively enroll 500 persons with chronic SCI (NParaplegia =250, NTetraplegia =250) in a web-based survey.
* Study participants will include males and females aged 18 years and older with SCI at the C5-L1 levels for more than 1 year.
* The investigators will consecutively enroll 75 persons with chronic tetraplegia aged 18 years and older with SCI at the C5-C8 levels for more than one year.
* The International Standards for Neurological Classification of SCI (ASIA/ISCoS)157 will serve as benchmarks for subject classification.
* A rater experienced in these procedures will classify study subjects.
* Persons from all ethnic and racial groups will be enrolled.
* The investigators will seek a gender distribution in proportion to population representation of persons with SCI (~80% male,

  ~20% female).
* After being provided with the study privacy practices, and HIPAA certification indicating available protections, participant candidates will undergo informed consent procedures approved by the Human Subjects Committee (IRB) at the University of Miami Miller School of Medicine (UM-MSOM).
* The investigators will consecutively enroll the first 25 persons from testing under Specific Aim 2 who satisfy criteria for diagnosis of SDB and consent to undergo additional study.

Exclusion Criteria:

* Subject candidates will be excluded for:

  1. previous diagnosis of SDB with active use of PAP,
  2. inability to read and comprehend English at a grade 5 level,
  3. requirement for day or night time non-invasive/invasive mechanical ventilation due to chronic respiratory failure,
  4. terminal illness in which life expectancy is less than one year,
  5. pregnancy,
  6. malignancy,
  7. surgery within 6 months,
  8. grade 2 or higher pressure ulcer within 3 months,
  9. recurrent acute infection or illness requiring hospitalization or IV antibiotics, and
  10. previous MI or cardiac surgery. The following medications and drug therapies will disqualify subjects from participating due to influences on lipids/lipoproteins, glucose/insulin, and inflammatory markers:
* lipid altering agents,
* β-adrenergic antagonists,
* maintenance α-blockers,
* insulin-sensitizers, and
* maintenance aspirin and
* non-steroidal anti-inflammatory drugs.

Blood sampling times will be altered in menstruating women to test during the follicular menstrual phase (cycle days 5-10), as recommended.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with Chronic Spinal Cord Injury who are asymptomatic for acute treable illness.
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To produce an evidence base for customary evaluation and treatment of SDB that will foster changes in medical practice patterns, while bringing attention to both SCI and their health providers of both apparent and obscure hazards of SDB. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States

REFERENCES:
- See also: Related Info — http://www.themiamiproject.org